CLINICAL TRIAL: NCT02807545
Title: Scoliosis-Specific Exercises for At-Risk Mild Adolescent Idiopathic Scoliosis Curves: A Multi-Site Preliminary Randomized Trial
Brief Title: Scoliosis-Specific Exercises for At-Risk AIS Curves
Acronym: EX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Collaborators: Scoliosis Research Society (Other); Boston Children's Hospital (Other); Columbia University (Other); Norton Leatherman Spine Center (Other); Johns Hopkins University (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Karina Zapata, PT, DPT, PhD, Principal Investigator, Texas Scottish Rite Hospital for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-15-1203
Record Dates: First submitted 2016-06-10; First posted 2016-06-21 (Estimated); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis-Specific Exercises; Schroth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Therapy Exercise Group (Experimental): Each patient assigned to the SSE group will attend at least 8 hours of supervised exercise training led by a Schroth-based certified physical therapist over the course of 6 months. Ideally, patients will be seen for 7 sessions.
  Patients will perform a home exercise program for 15 minutes a day, 5 days a week, when they can independently execute their prescribed exercises. An exercise log initialed by the guardian will help families keep track of their exercise adherence and serve as a way to monitor exercise adherence for patients who may not have a smartphone, tablet, or computer.
  Patients will also be able to meet with the therapists at their return-to-clinic visits and every 2-3 months thereafter until their 1 year follow-up to assess performance quality, maintain motivation, and progress intensity. Patients will be withdrawn if they do not achieve 80% exercise adherence within 6 months.
  Interventions: Behavioral: Scoliosis Specific Exercises
- Control Group (No Intervention): Patients randomized to this group will continue receiving standard-of-care treatment from their orthopaedic physician which includes regularly scheduled clinic visits and observation. Observation consists of no treatment of the scoliosis, only routine clinical assessment by the orthopaedic surgeon to detect curve progression every 3 to 6 months.

INTERVENTIONS:
Behavioral: Scoliosis Specific Exercises
  Other Names: Schroth-Based Method
  Arms: Physical Therapy Exercise Group

SUMMARY:
This study will be a multi-center, dual-arm randomized control study evaluating skeletally immature patients with mild AIS curves. At six institutions, patients will be randomized into either the scoliosis-specific exercise (SSE) treatment arm or a control group. The SSE group will receive training in SSE, posture, and activities of daily living by physical therapists certified in Schroth-based exercise methods. The control group will not receive SSE instruction and will only be observed by their treating orthopaedic surgeon (which is considered the standard-of-care treatment method). Results will be compared after one year of treatment.

DETAILED DESCRIPTION:
All patients with AIS meeting the following inclusion criteria will be eligible to participate in this trial: diagnosis of AIS; ages 10 to 17 years; major curve Cobb angles 15° to 20°; thoracolumbar, lumbar, or primary thoracic curve patterns; and Risser grade 0. Curves less than 15° will not be as clinically meaningful if they do not progress more than 5°. Curves 15° also allow for 5° of measurement error. Curves more than 20° will not be able to progress at least 5° before bracing is initiated according to SRS criteria (at 25°). Patients will be excluded according to the following exclusion criteria: scoliosis other than AIS, upper thoracic or double curve patterns, developmental disorders that prevent understanding and compliance with an exercise schedule, current or previous brace wear, and previous participation in a SSE program, previous spine surgery, inability to commit to performing a home exercise program for 15 minutes a day, 5 days a week, and inability to commit to attend at least 8 hours of PT within 6 months.

Patient medical records will be reviewed for eligibility. If a patient is deemed eligible for inclusion in the study, a member of the research team will meet with the patient and his or her family to review the consent form in a private medical exam room. The family will be given ample time to review the consent form and ask any questions. If a participant chooses to participate, a consent form will be signed by both the patient and the legal guardian prior to any investigational procedures occurring. Once a consent form has been signed, patients will be randomly assigned by the TSRH on site statistician to one of the two following groups:

1. Standardization of Physical Therapy:

   Physical therapists from Texas Scottish Rite Hospital, Boston Children's Hospital, Columbia University Medical Center, Norton Leatherman Spine Center, Johns Hopkins University, and Texas Children's Hospital who received training and certification in the Schroth-based (BSPTS) method have been recruited as members of the study team. Physical therapists at each institution will deliver a standardized exercise intervention.
2. Study Groups:

A) Scoliosis-Specific Exercise (SSE) Group

Each patient assigned to the SSE group will attend at least 8 hours of supervised exercise training led by a Schroth-based certified physical therapist over the course of 6 months. Ideally, patients will be seen for 7 sessions:

1. First session: 2 hours
2. Session 2: 1 hour (1 week later)
3. Session 3: 1 hour (1-2 weeks later)
4. Session 4: 1 hour (2-3 weeks after Session 3)
5. Session 5: 1 hour (3-4 weeks after Session 4)
6. Session 6: 1 hour (1-2 months after Session 5)
7. Session 7: 1 hour (1-2 months after Session 6)

The exact number of training sessions and time frame will be determined by the patient's ability to perform the exercises. All therapists will use a standardized exercise prescription algorithm and performance checklist similar to Dr. Parent's Schroth scoliosis exercise study. Patients will perform a home exercise program for 15 minutes a day, 5 days a week, when they can independently execute their prescribed exercises according to the following criteria:

1. Correctly move the pelvis so the body weight is over the base of support and neutral.
2. Accurately set up exercises per curve pattern in different positions. Exercises progress from static to dynamic and passive to active corrections.
3. Proficiently perform a minimum of 8 exercises integrating scoliosis-specific corrections which include auto-elongation to increase the spaces between the pelvis, vertebrae, and ribs. Various kinesthetic, mental imagery and proprioceptive strategies are used to further open concavities and depress convexities.
4. Perform scoliosis-specific corrections during activities of daily living. The overall goal is for patients to maintain a corrective posture throughout the day.

Patients will be asked to use a smartphone or tablet application (app) when performing the home exercise program which will be one method of tracking exercise adherence. A paper version of the app will be available to patients without access to a smartphone or tablet.

Patients will also be sent electronically a weekly survey regarding home exercise adherence through a secure research database, the Research Electronic Data Capture (REDCap). An exercise log initialed by the guardian will help families keep track of their exercise adherence and serve as a way to monitor exercise adherence for patients who may not have a smartphone, tablet, or computer.

Patients will also be able to meet with the therapists at their return-to-clinic visits and every 2-3 months thereafter until their 1 year follow-up to assess performance quality, maintain motivation, and progress intensity. Patients will be withdrawn if they do not achieve 80% exercise adherence within 6 months.

B) Control Group Patients randomized to this group will continue receiving standard-of-care treatment from their orthopaedic physician which includes regularly scheduled clinic visits and observation. Observation consists of no treatment of the scoliosis, only routine clinical assessment by the orthopaedic surgeon to detect curve progression every 3 to 6 months. Once all measurements have been collected at the patient's enrollment and one year followup, patients in this group will continue to be tracked through observation until skeletal maturity in order to record whether the patient experienced curve progression, was prescribed a brace, or proceeded to surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients diagnosed with Adolescent Idiopathic Scoliosis who meet the following inclusion criteria will be eligible to participate in this trial:

1. Age 10 to 17 years
2. Major curve Cobb angles of 12° to 24°
3. Risser Grade 0
4. Single thoracic, thoracolumbar, or lumbar curve patterns

Exclusion Criteria:

Patients will be excluded according to the following exclusion criteria:

1. Scoliosis other than AIS (congenital, neuromuscular, etc)
2. Upper thoracic or double curve patterns
3. Diagnosis of a developmental disorder that prevents understanding and compliance with an exercise schedule
4. Current or previous brace wear
5. Previous participation in a SSE program
6. Previous spine surgery
7. Patient inability to commit to attend at least 8 hours of PT within 6 months

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2023-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karina Zapata, PhD, Principal Investigator — Scottish Rite for Children
Locations (6):
- United States (6):
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Johns Hopkins, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
We never intended to make IPD available to other researchers. Our plan was only to share de-identified data with one lead institution.

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Therapy Exercise Group: Each patient assigned to the SSE group will attend at least 8 hours of supervised exercise training led by a Schroth-based certified physical therapist over the course of 6 months. Ideally, patients will be seen for 7 sessions.
  Patients will perform a home exercise program for 15 minutes a day, 5 days a week, when they can independently execute their prescribed exercises. An exercise log initialed by the guardian will help families keep track of their exercise adherence and serve as a way to monitor exercise adherence for patients who may not have a smartphone, tablet, or computer.
  Patients will also be able to meet with the therapists at their return-to-clinic visits and every 2-3 months thereafter until their 1 year follow-up to assess performance quality, maintain motivation, and progress intensity. Patients will be withdrawn if they do not achieve 80% exercise adherence within 6 months.
  Scoliosis Specific Exercises
Period: Overall Study
Arm/Group | Physical Therapy Exercise Group | Control Group
Started | 69 | 29
Completed (1 year follow-up) | 35 | 22 (1 year follow-up)
Not Completed | 34 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Therapy Exercise Group | Control Group | Total
Number analyzed (Participants) | 35 | 22 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 22 | 57
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (1.1) | 12.5 (1.4) | 11.9 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 15 | 41
  Male | 9 | 7 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 28 | 12 | 40
  Race/Ethnicity: Hispanic | 4 | 3 | 7
  Race/Ethnicity: Asian | 1 | 4 | 5
  Race/Ethnicity: African American | 1 | 1 | 2
  Race/Ethnicity: Native American | 1 | 1 | 2
  Race/Ethnicity: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 22 | 57
AIS Risser 0 curves 12-24 degrees [Mean (Standard Deviation); unit: degrees] | 16.2 (2.5) | 17.1 (2.9) | 16.6 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Overall Recruitment Rate
Description: Measured by the number of participants enrolled through study completion.
Time Frame: through study completion up to 45 months
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Therapy Exercise Group | Control Group
Number analyzed (Participants) | 69 | 29
Participants | 1 | 1

2. Primary Outcome: Treatment Attendance in the SSE Group
Description: Measured by the number of prescribed hours of physical therapy sessions attended after 1 year
Time Frame: after 1 year
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Physical Therapy Exercise Group
Number analyzed (Participants) | 35
hours | 9.7 (1.7)

3. Primary Outcome: Home Exercise Adherence in the SSE Group According to Weekly E-mails
Description: Measured by the percentage of prescribed exercises completed from baseline to 1 year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of exercises completed
Arm/Group | Physical Therapy Exercise Group
Number analyzed (Participants) | 35
percentage of exercises completed | 62.8 (37.8)

4. Secondary Outcome: Curve Magnitude
Description: Measured by the Cobb angle on radiograph
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Physical Therapy Exercise Group | Control Group
Number analyzed (Participants) | 35 | 22
degrees | 16.1 (7.1) | 18.1 (5.7)

5. Secondary Outcome: Curve Progression
Description: Percentage of participants whose curve progressed >5 degrees
Time Frame: after 1 year
Population: Out of the 35 participants in the Exercise group who completed the study and 22 participants in the Control group who completed the study, 34 participants in the Exercise group and 21 participants in the Control group had curve magnitude data to report curve progression, since 1 patient in each group did not receive radiographic measurements at that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Therapy Exercise Group | Control Group
Number analyzed (Participants) | 34 | 21
Participants | 8 | 7

6. Secondary Outcome: Brace Prescription
Description: Measured by the percentage of participants prescribed a brace
Time Frame: after 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Physical Therapy Exercise Group | Control Group
Number analyzed (Participants) | 35 | 22
Participants | 9 | 12

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Physical Therapy Exercise Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/22
Other Adverse Events (participants affected / at risk) | 0/35 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT02807545/Prot_SAP_000.pdf